CLINICAL TRIAL: NCT07368361
Title: "Comparative Outcomes of Mucosal Reset (Reboot) Versus Complete Sinusotomy (Full House FESS) in CRSwNP: A Prospective Study
Brief Title: Th Study Wants to Compare the Best Technique for Sinus Operation in CRSWNP
Acronym: REBOOT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kafrelsheikh University (Other)
Responsible Party: Principal Investigator, Amr Mahr Shady, resident, Kafrelsheikh University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KFSIRB200-710
Record Dates: First submitted 2025-12-25; First posted 2026-01-26 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2025-12

CONDITIONS: CRSWNP
Keywords: REBOOT, SINUSOTOMY, FULL HOUSE FESS, CRSWNP

STUDY DESIGN:
Intervention Model Description: This randomized controlled trial aims to compare the efficacy and safety of reboot surgery versus conventional full house FESS in patients with refractory CRSwNP
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- "Comparative Outcomes of Mucosal Reset (Reboot) IN CRSWNP (Experimental): The first group will undergo Reboot operation" Complete removal of inflamed mucosa to periosteum"
  Interventions: Device: Reboot operation" Complete removal of inflamed mucosa to periosteum"
- Complete Sinusotomy (Full House FESS IN CRSWNP (Experimental): the second group will have a conventional FESS operation " Mucosal preservation where healthy"
  Interventions: Device: endoscopic nasal operation

INTERVENTIONS:
Device: endoscopic nasal operation — . conventional FESS operation "
  Arms: Complete Sinusotomy (Full House FESS IN CRSWNP
Device: Reboot operation" Complete removal of inflamed mucosa to periosteum" — Reboot operation" Complete removal of inflamed mucosa to periosteum"
  Arms: "Comparative Outcomes of Mucosal Reset (Reboot) IN CRSWNP

SUMMARY:
This randomized controlled trial aims to compare the efficacy and safety of reboot surgery versus conventional full house FESS in patients with refractory CRSwNP, focusing on:

1. Primary Outcome:

* Compare 24-month recurrence rates (defined as endoscopic polyp score ≥2) 2. Secondary Outcomes:
* Recurrence-free survival (time to first recurrence), Quality of life improvement (SNOT-22 scores), Reduction in systemic corticosteroid use, Complication rates (synechiae, bleeding, infection) and Cost-effectiveness of each approach

DETAILED DESCRIPTION:
Chronic Rhinosinusitis (CRS) affects 5-15% of people globallymmmmm. Traditionally classified as with polyps (CRSwNP) or without (CRSsNP), modern approaches now focus on endotype-based categorization.CRSwNP, linked to type-2 inflammation[4], often causes severe, recurrent symptoms that significantly impair quality of life and increase healthcare costs.[5] Despite this, its impact is frequently underestimated, leading to improper treatment-such as overuse of oral steroids-which risks long-term side effects.

Effective control often requires multimodal therapy, yet results remain inconsistent. Recently, monoclonal antibodies (mAbs) targeting type-2 inflammation have revolutionized treatment, offering long-term relief and addressing comorbidities.

Despite these advances, surgery-particularly endoscopic sinus surgery (ESS)-remains pivotal, especially as initial therapy. ESS continues to evolve, balancing effectiveness, invasiveness, and cost.

For refractory CRSwNP with rapid post-surgery recurrence, repeated interventions are often needed. Recent strategies like the "reboot approach"-complete removal of inflamed sinus mucosa down to the bone-aim to reset the inflammatory environment and promote healthier mucosal regeneration (Alsharif et al.) .

The aim here is to demonstrate how effectiveness of "Reboot surgery: for chronic sinusitis with polyps reduces recurrences, extends symptom-free periods, improves quality of life, and decreases steroid use. We analyze its benefits and limitations based on type 2 inflammation mechanisms.

ELIGIBILITY:
Inclusion Criteria:Patients above the age of 18 years presenting with recurrent refractory CRSwNP (failed ≥1 biologic/prior FESS), Type-2 endotype confirmation (blood/tissue eosinophilia, IgE ≥100 IU/mL), Lund-Mackay CT score ≥10 will be included in the study.

Exclusion Criteria:

eosinophilic granulomatosis with polyangiitis (EGPA) or severe systemic diseases (except controlled asthma or NSAID-exacerbated respiratory disease), neoplasms, vasoconstrictor abuse (e.g., oxymetazoline dependence), unilateral nasal inflammatory disease, bilateral inflammatory disease without polyps, or treatment with monoclonal antibodies in the past 12 months, Patients younger than 18 years of age and patients are unfit for general anesthesia.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
"Comparative Outcomes of Mucosal Reset (Reboot) Versus Complete Sinusotomy (Full House FESS) in CRSwNP: A Prospective Study | 1-1-2027
  24-month recurrence rates (defined as endoscopic polyp score ≥2)

CONTACTS AND LOCATIONS:
Locations (1):
- Kafrelsheikh Faculty of Medicine, Egypt, Kafrelsheikh, Canada

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Fokkens WJ, Lund VJ, Hopkins C, Hellings PW, Kern R, Reitsma S, Toppila-Salmi S, Bernal-Sprekelsen M, Mullol J, Alobid I, Terezinha Anselmo-Lima W, Bachert C, Baroody F, von Buchwald C, Cervin A, Cohen N, Constantinidis J, De Gabory L, Desrosiers M, Diamant Z, Douglas RG, Gevaert PH, Hafner A, Harvey RJ, Joos GF, Kalogjera L, Knill A, Kocks JH, Landis BN, Limpens J, Lebeer S, Lourenco O, Meco C, Matricardi PM, O'Mahony L, Philpott CM, Ryan D, Schlosser R, Senior B, Smith TL, Teeling T, Tomazic PV, Wang DY, Wang D, Zhang L, Agius AM, Ahlstrom-Emanuelsson C, Alabri R, Albu S, Alhabash S, Aleksic A, Aloulah M, Al-Qudah M, Alsaleh S, Baban MA, Baudoin T, Balvers T, Battaglia P, Bedoya JD, Beule A, Bofares KM, Braverman I, Brozek-Madry E, Richard B, Callejas C, Carrie S, Caulley L, Chussi D, de Corso E, Coste A, El Hadi U, Elfarouk A, Eloy PH, Farrokhi S, Felisati G, Ferrari MD, Fishchuk R, Grayson W, Goncalves PM, Grdinic B, Grgic V, Hamizan AW, Heinichen JV, Husain S, Ping TI, Ivaska J, Jakimovska F, Jovancevic L, Kakande E, Kamel R, Karpischenko S, Kariyawasam HH, Kawauchi H, Kjeldsen A, Klimek L, Krzeski A, Kopacheva Barsova G, Kim SW, Lal D, Letort JJ, Lopatin A, Mahdjoubi A, Mesbahi A, Netkovski J, Nyenbue Tshipukane D, Obando-Valverde A, Okano M, Onerci M, Ong YK, Orlandi R, Otori N, Ouennoughy K, Ozkan M, Peric A, Plzak J, Prokopakis E, Prepageran N, Psaltis A, Pugin B, Raftopulos M, Rombaux P, Riechelmann H, Sahtout S, Sarafoleanu CC, Searyoh K, Rhee CS, Shi J, Shkoukani M, Shukuryan AK, Sicak M, Smyth D, Sindvongs K, Soklic Kosak T, Stjarne P, Sutikno B, Steinsvag S, Tantilipikorn P, Thanaviratananich S, Tran T, Urbancic J, Valiulius A, Vasquez de Aparicio C, Vicheva D, Virkkula PM, Vicente G, Voegels R, Wagenmann MM, Wardani RS, Welge-Lussen A, Witterick I, Wright E, Zabolotniy D, Zsolt B, Zwetsloot CP. European Position Paper on Rhinosinusitis and Nasal Polyps 2020. Rhinology. 2020 Feb 20;58(Suppl S29):1-464. doi: 10.4193/Rhin20.600. PMID 32077450
- [Result] Alsharif S, Jonstam K, van Zele T, Gevaert P, Holtappels G, Bachert C. Endoscopic Sinus Surgery for Type-2 CRS wNP: An Endotype-Based Retrospective Study. Laryngoscope. 2019 Jun;129(6):1286-1292. doi: 10.1002/lary.27815. Epub 2019 Jan 21. PMID 30663058